CLINICAL TRIAL: NCT03514784
Title: Road to Discovery for Combination Probiotic BB-12 With LGG (Different Doses) in Treating Autism Spectrum Disorder Disorders
Brief Title: Combination Probiotic: BB-12 With LGG (Different Doses) in Treating Children With Autism Spectrum Disorder
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Texas Higher Education Coordinating Board (Other Government); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, J. Marc Rhoads, Director, Pediatric Gastroenterology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-17-0995; R01HD095158-02 (NIH); NCT02674984 (obsolete NCT alias)
Record Dates: First submitted 2018-01-26; First posted 2018-05-02 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Autism Spectrum Disorder; Gastrointestinal Symptoms
Keywords: Autism Spectrum Disorder, ASD, Gastrointestinal Symptoms, Constipation, Diarrhea
MeSH Terms: conditions — Autism Spectrum Disorder; Constipation; Diarrhea | interventions — Probiotics; maltodextrin

STUDY DESIGN:
Intervention Model Description: After psychological screening, the subjects will be randomize children to one of 3 groups. The total number of subject to be enrolled will be 70 healthy children with confirmed ASD status, randomizing each child to placebo (maltodextrin), low daily dose (1 billion cfu's), and higher daily dose (10 billion cfu's) of BB-12+LGG once daily at 1:2:2 ratio. Data will be combined with 30 patients obtained from two funding sources: Texas (THECB) and U.T. pilot project. The data will be combined and an identical design of the placebo and 1 billion cfu dose arms.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The head statistician and study pharmacist will be aware of randomization scheme. The investigators will use an adaptive minimization program for randomization that balances the 3 study arms with respect to distributions of sex and age (4-10 vs. 11-16 y.o.). Patients will be randomized to placebo, 1 billion CFU, and 10 billion CFU study arms at a ratio of 1:2:2. (Currently marketed over-the-counter probiotics typically contain 0.1-50 billion CFUs per dose.) The performance of our covariate adaptive randomization algorithm will be verified through simulation studies before implementation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BB-12 with LGG (Lower Dose) (Active Comparator): BB-12 with LGG (Multistrain probiotic; lower dose): 1 billion CFUs
  Interventions: Drug: BB-12 with LGG (Lower Dose)
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Drug: Placebo
- BB-12 with LGG (Higher Dose) (Active Comparator): BB-12 with LGG (Multistrain probiotic: higher dose): 10 billion CFUs
  Interventions: Drug: BB-12 with LGG (Higher Dose)

INTERVENTIONS:
Drug: BB-12 with LGG (Higher Dose) — BB-12 with LGG - Higher Dose (10 billion CFUs)
  Other Names: Probiotic
  Arms: BB-12 with LGG (Higher Dose)
Drug: Placebo — Maltodextrin
  Other Names: Maltodextrin
  Arms: Placebo
Drug: BB-12 with LGG (Lower Dose) — BB-12 with LGG - Lower Dose (1 billion CFUs)
  Other Names: Probiotic
  Arms: BB-12 with LGG (Lower Dose)

SUMMARY:
This protocol is a blinded randomized controlled study of the effects of BB-12 with LGG at different doses in 70 healthy children with autism spectrum disorders at lower and higher doses over an 56-day period and a 28- day observation period. The study is being conducted in order to assess safety and tolerability of the probiotic (BB-12 with LGG) at 2 different doses of BB-12 with LGG. Identifying effects on behaviors in healthy children with ASD using SRS-2 and ABC, GI symptoms using GI symptom severity index, and relevant biomarkers of inflammation, microbiota, and metabolites. Primary testing and procedures will be conducted at the University of Texas Health Science Center at Houston and Memorial Hermann.

Biomarker identification includes Integrative analysis of plasma metabolome and stool microbiota will be conducted with the collaboration of Dr. Ruth Ann Luna and Dr. Jim Versalovic at Alkek Center for Metagenomics and Microbiome Research, Department of Molecular Virology & Microbiology of Baylor College of Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children with autism spectrum disorders (4 - 16 years old) and gastrointestinal symptoms, based on the GI Severity Index, with no other recognized illness will be enrolled in this study. There will be no selection on the basis of age, race, or gender. Although the investigators anticipate the majority of subjects will be male and/or pre-pubertal, in females of childbearing potential, a pregnancy test (urine) will be performed on females participating (at each visit).

Exclusion Criteria:

* Pregnancy or breastfeeding
* Subjects taking immunosuppressive medications, including oral corticosteroids
* A History of Positive result of HIV, Hepatitis B, and/or Hepatitis C test
* Abnormal lab test results (Section 5.2)
* Gastrointestinal diseases such as celiac disease, inflammatory bowel disease
* Subjects with an allergy to antibiotics
* Presence of fever or a pre-existing adverse event monitored in the study
* Use of probiotics in the last 30 days
* Acute diarrheal illness within the past 30 days
* Recent (within 2 weeks) or current use of oral antibiotics /anti-fungals Current use of oral laxatives
* Subjects with implanted prosthetic devices including prosthetic heart valves
* The investigators will require that subject not take any other probiotic-containing products, including yogurt supplemented with probiotics during the study period.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Effects of BB-12+LGG at different doses on adverse events (safety) | 84 days
  Adverse events (Safety) will be measured by case report form (survey) that are related to BB-12 with LGG (health-promoting bacteria) or placebo treatment. The symptom grade will detail the severity of adverse events.

SECONDARY OUTCOMES:
Effects of BB-12+LGG at different doses on irritability and maladaptive behaviors with Aberrant Behavior Checklist (ABC) | Days 1, 21, 56 and 84
  Psychological/Behavioral change in irritability and related maladaptive behaviors associated with ASD will be measured by the Aberrant Behavior Checklist (ABC) pre and post treatment
Effects of BB-12+LGG at different doses on irritability and maladaptive behaviors measured with the Social Responsiveness Scale-2 | Days 1, 21, 56 and 84
  Psychological/Behavioral change in irritability and related maladaptive behaviors associated with ASD will be measured by the and the Social Responsiveness Scale-2 (SRS-2) pre and post treatment.

OTHER OUTCOMES:
Effects of BB-12+LGG at different doses on GI symptoms as measured by GI Symptom Severity Index | Days 1, 21, 56 and 84
  GI symptoms will be measured by the GI Severity Index.
Effects of BB-12+LGG at different doses on gut inflammation (S1009A) | Days 1, 56 and 84
  Plasma S100A9 will indicate GI and systemic levels of inflammation. S100A9 is a damage-associated molecular pattern molecule (DAMP) released by granulocytes, which is reportedly elevated 2-fold in plasma of children with ASD.
Effects of BB-12+LGG at different doses on gut inflammation (Fecal Calprotectin) | Days 1, 56 and 84
  Biological change in fecal calprotectin levels. FC is a highly accurate fecal marker of inflammation.
Effects of BB-12+LGG at different doses on gut inflammation (Plasma Zonulin) | Days 1, 56 and 84
  Plasma zonulin, a marker for intestinal permeability ("leaky gut"), which is often associated with inflammation.
Effects of BB-12+LGG at different doses on gut inflammation (IL-8) | Days 1, 56 and 84
  IL-8 can be an indicator of gut inflammation; it released from the intestinal epithelial cells during inflammation.
Effects of BB-12+LGG at different doses on fecal microbial community | Days 1, 56 and 84
  Using 16S rDNA analysis, this will determine microbial alpha and beta diversity and distribution of the major taxa before and after probiotic treatment.
Effects of BB-12+LGG at different doses on metabolites | Days 1, 56 and 84
  This will determine levels of metabolic markers which are reported to be abnormal in autism: fecal amino acids, ammonia, short chain fatty acids (SCFA), and phenols.

CONTACTS AND LOCATIONS:
Overall Officials: J Marc RHoads, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- UTHealth, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No